CLINICAL TRIAL: NCT05062941
Title: The Effect of High-intensity Laser Therapy on Pain, Functionality, and Quality of Life in Patients With Chronic Shoulder Pain
Brief Title: The Effect of High-intensity Laser Therapy in Patients With Chronic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28.03.2018.217
Record Dates: First submitted 2021-09-09; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Chronic Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Conventional therapy (CT) was applied to all participants. CT included application of 15 minutes of hot-pack, 20 minutes of transcutaneous electrical nerve stimulation (TENS) in conventional mode, 5 minutes of ultrasound (1.5 W/cm2, 1 MHz), 20 minutes of interference current with vacuum electrodes (80 Hz pulse frequency, 1/1 rectangular spectrum), and exercises (all exercises were applied as 1 set of 10 repetitions in each direction: Codman exercises (3-directions), wand exercises (4-directions), exercises using the shoulder wheel (2-directions), exercises with exercise band (5-directions), exercises on the finger ladder (1 set of 10 repetitions in both directions); and shoulder capsule stretching exercises performed (1 set of 12 repetitions) by asking the subjects to wait 20 seconds where the tension was felt).
  Interventions: Other: Conventional physiotherapy
- Study group (Active Comparator): Same conventional therapy (CT) that was applied to control group was also applied to all participants in this group. CT included application of 15 minutes of hot-pack, 20 minutes of transcutaneous electrical nerve stimulation (TENS), 5 minutes of ultrasound, 20 minutes of interference current with vacuum electrodes, and the same exercises.
  In addition to the CT program, only study group has received HILT (BTL 6000, BTL Industries, Inc., USA) application to the shoulder area (analgesic mode, 25 Hz,10 W, 12 j/cm2) for 2 minutes.
  Interventions: Other: Conventional physiotherapy; Device: High-intensity laser therapy (HILT)

INTERVENTIONS:
Other: Conventional physiotherapy — Conventional therapy (CT) included application of 15 minutes of hot-pack, 20 minutes of transcutaneous electrical nerve stimulation, 5 minutes of ultrasound, 20 minutes of interference current with vacuum electrodes, and exercises.
Device: High-intensity laser therapy (HILT) — HILT stimulates oxidation of mitochondria and ATP creation by delivering high energy output inside the tissues and with this photochemistry effect, metabolism and blood circulation is increased resulting HILT to cause quick absorption of edema and removal of exudates.
  HILT (BTL 6000, BTL Industries, Inc., USA) application was to the shoulder area in the analgesic mode of the device at a frequency of 25 Hz with a power of 10 W and a dosage of 12 j/cm2 for 2 minutes: 5 sessions a week for 3 weeks and 15 sessions in total.
  Arms: Study group

SUMMARY:
The aim of this study was to investigate the effects of biostimulating, analgesic and noninvasive high intensity laser therapy on pain, functionality and quality of life in patients with chronic shoulder pain. Participants between the ages of 18-75 and without any cognitive, communication and psychiatric problems were included in the study. Patients were randomized into two groups and both received conventional physiotherapy and rehabilitation program for 3 weeks, 5 sessions a week. The treatment program applied was as followed; the control Group (n = 25): conventional physiotherapy and study Group (n = 25): conventional physiotherapy and High-intensity Laser Therapy (HILT). Upper extremity range of motion was evaluated with 'goniometer', pain threshold with 'algometer, muscle strength with 'myometer'; disability status with 'The Disabilities of the Arm, Shoulder and Hand (DASH)'.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of biostimulating, analgesic and noninvasive high intensity laser therapy on pain, functionality and quality of life in patients with chronic shoulder pain. Participants between the ages of 18-75 and without any cognitive, communication and psychiatric problems were included in the study. Patients were randomized into two groups and both received conventional physiotherapy and rehabilitation program for 3 weeks, 5 sessions a week. The treatment program applied was as followed; the control Group (n = 25): conventional physiotherapy and study Group (n = 25): conventional physiotherapy and High-intensity Laser Therapy (HILT). Upper extremity range of motion was evaluated with 'goniometer', pain threshold with 'algometer, muscle strength with 'myometer'; disability status with 'The Disabilities of the Arm, Shoulder and Hand (DASH)'.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in the study,
* Aged 18-75 years
* being diagnosed with chronic shoulder pain

Exclusion Criteria:

* not having sufficient cooperation to follow exercises,
* having any communication problems or psychiatric problems,
* having any cardiac or orthopedic discomfort that may prevent the application of evaluation methods.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in range of motion from baseline to week 3 | 3 weeks
  The range of motion of the joints in the upper extremities will be measured using the universal goniometer before and after the treatment.
Change in pain threshold from baseline to week 3 | 3 weeks
  The pain threshold will be measured with a digital algometer device. Algometers are devices that can be used to identify the pressure and/or force eliciting a pressure-pain threshold. It has been noted in pressure-pain threshold studies that the rate at which manual force is applied should be consistent to provide the greatest reliability.
Change in disability of the upper extremity from baseline to week 3 | 3 weeks
  Disability of the upper extremities will be assessed with 'The Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire'. It is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The questionnaire was designed to help describe the disability experienced by people with upper-limb disorders and also to monitor changes in symptoms and function over time. The 30-item questionnaire includes 21 physical function items, 6 symptom items, and 3 social/role function items. Each 30 items are marked from 1 (No Difficulty) to 5 (Unable). DASH are added to form the raw, or actual, score. A minimum score is 30; a maximum is 150. The range of the scores, therefore-from 30 to 150-equals 120. The raw score is then transformed to a zero-to-100 scale with zero reflecting no disability (good function) and 100 reflecting maximum disability.
Change in muscle strength from baseline to week 3 | 3 weeks
  The muscle strength of shoulder flexion, abduction, adduction, external and internal rotation movements will be evaluated by using the Baseline Push-Pull (New York) dynamometer. Results will be calculated in kg (1 lb = 0.454 kg). The patient's arm will be stabilized and the patient will be asked to show maximum resistance within 2 sec against the dynamometer placed and then hold it for 5 seconds at this position and power. The measurement will be repeated twice and recorded with the average of these two values.
Change in health status from baseline to week 3 | 3 weeks
  In the evaluation of the health status of the individuals the Short Form-36 (SF-36) questionnaire was used. SF-36 is a questionnaire developed to self-evaluate the quality of life. It consists of 36 items in total and has eight sub-parameters. Subscales are scored between 0 and 100, and higher scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zubeyir Sari, Prof., Study Director — Marmara University
Locations (1):
- Cadde Medical Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No